CLINICAL TRIAL: NCT03575988
Title: Department of Solemn Scientific Research Platform in Liaoning University of Traditional Chinese Medicine
Brief Title: Early Changes in Pulmonary Function and Vascular Endothelial Function and the Correlation Between Them in T2DM Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guanlin Yang (Other)
Responsible Party: Sponsor-Investigator, Guanlin Yang, Guan-lin Yang is the presidentg and full Clinical professor(Cardiovascular medicine) of Liaoning University of Traditional Chinese Medicine, Liaoning University of Traditional Chinese Medicine
Organization: Liaoning University of Traditional Chinese Medicine (Other)
Other Study IDs: 2018052802
Record Dates: First submitted 2018-06-02; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Pulmonary function; Vascular endothelial function; Ultrasound
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes group
  Interventions: Other: Diabetes
- Control group
  Interventions: Other: Diabetes

INTERVENTIONS:
Other: Diabetes — The patients have diabetes without diabetic retinopathy from the diabetic outpatient

SUMMARY:
Current knowledge: To the best of our knowledge, no studies have reported the correlation between pulmonary function and the vascular endothelial function in diabetic patients during the preclinical period. Indeed, diabetic nephropathy and retinopathy are the leading causes of end-stage renal failure and acquired blindness, respectively. However, when investigators treat patients with type 2 diabetes, investigators seldom consider the pulmonary vascular injury induced by glycemia. Experimental studies have shown that pulmonary function and Vascular endothelial function change during the preclinical stages of diabetic retinopathy. Researchers have already established that compared to healthy subjects, patients with type 2 diabetes have a reduced alveolar gas exchange capacity. The NO and ET-1 can be used to assess the Vascular endothelial function.

What this paper contributes to our knowledge: Regulating glycemia can improve Vascular endothelial function . This study suggests that detecting the NO and ET-1 would allow for the prediction of changes in pulmonary function during the preclinical stages of diabetic retinopathy and the degree of retinopathy in the future.

ELIGIBILITY:
Inclusion Criteria:1) symptoms of diabetes (thirst, polydipsia, diuresis, and unexplainable weight loss); 2) random blood sugar ≥11.1 mol/L, fasting plasma glucose ≥7.0 mol/L or an oral glucose tolerance test outcome (2-hour postprandial blood glucose) ≥11.1 mol/L; or 3) no symptoms of diabetes but either random blood sugar ≥11.1 mol/L or fasting plasma glucose ≥7.0 mol/L.

-

Exclusion Criteria:1) diagnosis of type 2 diabetes according to the guidelines of the American Diabetes Association;11 2) no history of smoking (never smoked), pulmonary disease or pulmonary infection (during the treatment or recovery period); 3) no hepatopathy, nephropathy, or gastrointestinal disease; and 4) a high likelihood of good compliance and the ability to visit our hospital for periodic assessments. The exclusion criteria were as follows: 1) diagnosis of type 1 diabetes; 2) pregnancy and/or active lactation; 3) intensive care with insulin treatment; 4) renal inadequacy, hypohepatia, or heart disease; 5) pneumonia, influenza (during the treatment or recovery period), phthisis or other pulmonary infection; 6) presence of multiple pulmonary cysts, bullae of the lung, or diffuse pulmonary calcifications confirmed via CT; 7) combined diabetic retinopathy and hypertension (for which antihypertensive drugs are used); 8) aneurysm, dissection of aorta; 9) inadequate control of serum lipid parameters by cholesterol-lowering drugs; 10) body mass index ≥32; and 11) the use of systemically injected glucocorticoids within 3 months prior to our study.

-

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The diabetes duration (range 3 to 12 years), body mass index (range 23 to 31 kg/m2), glycosylated hemoglobin A1c levels [range 7.0% (53 mmol/mol) to 10% (86 mmol/mol)], pulmonary function parameters, retrobulbar hemodynamic parameters (bilateral resistivity index), serum lipid parameters (i.e., total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and triglyceride), and blood pressure were recorded
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-07-03 (Estimated); Primary Completion 2018-11-03 (Estimated); Study Completion 2019-06-03 (Estimated)

PRIMARY OUTCOMES:
pulmonary function parameters(vital capacity,VC,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(forced vital capacity,FVC,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(forced expiratory volume in 1 second,FEV1,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(peak expiratory force,PEF,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(maximal voluntary ventilation,MVV,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(total lung capacity,TLC,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(forced expiratory volume in 1 second/ forced vital capacity,FEV1/FVC,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(diffusing capacity for carbon monoxide of lung,DLCO,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.
pulmonary function parameters(diffusing capacity for carbon monoxide of lung/unit volume,DLCO/VA,%) | one week
  Pulmonary function tests were performed using a spirometer. We used the ratio of measured values to the expected values, % of predicted value, to eliminate the influence of age, height, and weight. Before testing, subjects remained sitting at quiet rest for at least 30 min, pulmonary function tests were performed 3 times and the best of 3 acceptable readings was used in the analysis. Spirometry and analysis of pulmonary function were performed by trained professionals.

SECONDARY OUTCOMES:
Vascular endothelial function(nitrogen oxide,NO,μmol /L) | one week
  NO were detected by biochemical radioimmunoassay (biochemical,μmol /L),ET-1(radioimmunoassay,μg /L) were dectcted in sugar
Vascular endothelial function(endothelin-1,ET-1,μmol /L) | one week
  ET-1 were detected by biochemical radioimmunoassay

OTHER OUTCOMES:
Blood sugar(2-hour postprandial blood glucose , 2hPBG(mmol/l)) | one week
  Plasma glucose levels were determined by the glucose oxidase method. The OGTT method used 75 g of oral glucose (50% anhydrous glucose solution 150 ml including 7.5 bottles added to 150 ml warm water). Venous blood was extracted to measure the 2hPG, and 5 ml of venous blood was placed into a glass tube, left standing at least 10 min, and centrifuged (3000 r/min) 10 min to separate serum, which was saved in -70 ℃ cryogenic refrigerator
Blood sugar(fasting plasma glucose,FPG(mmol/l)) | one week
  Plasma glucose levels were determined by the glucose oxidase method. The OGTT method used 75 g of oral glucose (50% anhydrous glucose solution 150 ml including 7.5 bottles added to 150 ml warm water). Venous blood was extracted to measure the 2hPG, and 5 ml of venous blood was placed into a glass tube, left standing at least 10 min, and centrifuged (3000 r/min) 10 min to separate serum, which was saved in -70 ℃ cryogenic refrigerator
Blood sugar(glycosylated hemoglobinA1c,HbA1c(%)) | one week
  Plasma glucose levels were determined by the glucose oxidase method. The OGTT method used 75 g of oral glucose (50% anhydrous glucose solution 150 ml including 7.5 bottles added to 150 ml warm water). Venous blood was extracted to measure the 2hPG, and 5 ml of venous blood was placed into a glass tube, left standing at least 10 min, and centrifuged (3000 r/min) 10 min to separate serum, which was saved in -70 ℃ cryogenic refrigerator
Serum lipid(Total cholesterol,TC(mg/dl)) | on week
  TC were measured according to the research kit instructions. All the specimens were measured within 1 week of collection.
Serum lipid(High-density lipoprotein cholesterol,HDL-C(mg/dl)) | on week
  HDL-C were measured according to the research kit instructions. All the specimens were measured within 1 week of collection.
Serum lipid(Low-density lipoprotein cholesterol,LDL-C(mg/dl)) | on week
  LDL-C were measured according to the research kit instructions. All the specimens were measured within 1 week of collection.
Serum lipid(Triglycerides,TG(mg/dl)) | on week
  TG were measured according to the research kit instructions. All the specimens were measured within 1 week of collection.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tai H, Jiang XL, Yao SC, Liu Y, Wei H, Li LB, Jiao ZJ, Wang TQ, Kuang JS, Jia LQ. Vascular Endothelial Function as a Valid Predictor of Variations in Pulmonary Function in T2DM Patients Without Related Complications. Front Endocrinol (Lausanne). 2021 Mar 11;12:622768. doi: 10.3389/fendo.2021.622768. eCollection 2021. PMID 33776922